CLINICAL TRIAL: NCT04115124
Title: The Efficacy of Ethnographic Participatory Action Research In Decreasing the Incidence of Female Genital Mutilation in Nigeria
Brief Title: Using Ethnographic Participatory Action Research to Decrease the Incidence of Female Genital Mutilation in Nigeria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lifespan Healthcare Resource Limited (Other)
Responsible Party: Principal Investigator, Dr.Ihedioha Emmanuel Chukwunwike, Principal Investigator, Lifespan Healthcare Resource Limited
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ST-POC-1908-25739
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Behavior, Social
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-PAR Arm (Experimental): Exposed to media, information and communication technology through ethnographic participatory action research.
  Interventions: Behavioral: Participatory Action Research

INTERVENTIONS:
Behavioral: Participatory Action Research — The research will employ a Participatory Action research quasi-experimental pre-post test study design .

SUMMARY:
Female Genital Mutilation(FGM) is a harmful practice on girls and women which causes irreparable sexual, reproductive and psychological harm. It is an act of violence, extreme discrimination and fundamental human rights violation against women and girls. This practice leaves victims feeling scared, psychologically scarred and distressed. FGM sustains deep rooted inequality between the sexes, constitutes a barrier to female civic participation and social inclusion and therefore, leads to inequitable socio- economic growth and prosperity. The World Health Organization(WHO) estimates that an alarming 200 million girls alive today have undergone FGM, while an estimated 3 million girls are at risk annually. A common factor influencing the continuation of FGM is the need to conform to social norms. Social norms among other roles, influence behaviors that shape people's ability to protect their health and achieve their life potential.

Methods: The investigators have designed a quasi-experimental comparison group pre-post test study involving members of Oduma, Okigwe, Nkerefi, Edda communities in Eastern Nigeria. Our study will run for a period of 12 months. The investigators expect that the outcome of this study will lead to policy changes placing emphasis on using participatory action research in addressing FGM in Nigeria.

DETAILED DESCRIPTION:
FGM is a harmful practice on girls and women which causes irreparable sexual, reproductive and psychological harm. It is an act of violence, extreme discrimination and fundamental human rights violation against women and girls. This practice leaves victims feeling scared, psychologically scarred and distressed. FGM sustains deep rooted inequality between the sexes, constitutes a barrier to female civic participation and social inclusion and therefore, leads to inequitable socio- economic growth and prosperity. The WHO estimates that an alarming 200 million girls alive today have undergone FGM, while an estimated 3 million girls are at risk annually. A common factor influencing the continuation of FGM is the need to conform to social norms. Social norms among other roles, influence behaviors that shape people's ability to protect their health and achieve their life potential.

Methods: The investigators have designed a quasi-experimental comparison group pre-post test study involving members of Oduma community in Ebonyi state. This research study will run for a period of 12 months. The investigators expect that the outcome of this study will lead to policy changes placing emphasis on using participatory action research in addressing FGM in Nigeria

Rationale There is a considerable lack of information on the efficacy of interventions to reduce the prevalence of FGM in Nigeria. In addition, this research study is needed to provide critical updated information on the efficacy of participatory action research in improving communities knowledge and attitude towards SHRH and how this affects the prevalence of FGM.

Objectives:

To determine the efficacy of e- PAR in reducing the incidence of FGM in Nigeria.

To determine the efficacy of e-PAR in improving Sexual Reproductive Health and Rights(SRHR) knowledge.

To determine the efficacy of e-PAR in improving Sexual Reproductive Health and Rights (SRHR) attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Consenting Participants living in the intervention communities.
* Consenting community health workers working in the intervention communities.
* Consenting patent medicine sellers working in the intervention communities.

Exclusion Criteria:

-

Ages: 1 Year to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Female Genital mutilation Secondary to Ethnographic Participatory Action Research(PAR) Intervention. | 12 months
  Number of Cut Girls secondary to PAR Intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Ihedioha, MD, Principal Investigator — Lifespan Heathcare Resource
Locations (1):
- Oduma, Oduma, Ebonyi State, Nigeria